CLINICAL TRIAL: NCT01594411
Title: Investigation of a Molecular Personalized Coronary Gene Expression Test (Corus CAD or ASGES) on Primary Care Practice Pattern
Brief Title: PCP Use of a Gene Expression Test (Corus CAD or ASGES) in Coronary Artery Disease Diagnosis
Acronym: IMPACT-PCP
Status: Completed | Type: Observational
Sponsor: CardioDx (Industry)
Responsible Party: Sponsor
Other Study IDs: CDX_000014; IMPACT-PCP (Other: CardioDx)
Record Dates: First submitted 2012-04-20; First posted 2012-05-09 (Estimated); Results first posted 2014-04-23 (Estimated); Last update posted 2019-01-31 (Actual); Status verified 2019-01

CONDITIONS: Chest Pain; Cardiovascular Diseases; Angina Pectoris; Coronary Artery Disease; CAD; CVD; CHD; Coronary Heart Disease
Keywords: Corus CAD; ASGES; Age/Sex/Gene Expression Score; Gene Expression; GES; CAD; CVD; CHD; Clinical Utility; Precision Medicine; Primary care; Coronary Artery Disease; Angina Pectoris; Chest Pain; Cardiovascular Disease; Coronary Heart Disease; IMPACT; IMPACT-PCP
MeSH Terms: conditions — Chest Pain; Cardiovascular Diseases; Angina Pectoris; Coronary Artery Disease; Coronary Disease; Tooth, Impacted

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — One 2.5 mL PAXgene (PreAnalytiXTM) (for RNA preservation) tube will be filled with approximately 7.5 ml of blood and sent to CardioDx, Inc. for analysis.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- All subjects: Subjects are enrolled at multiple participating primary care practices. The main inclusion criterion for enrollment is the occurrence of chest pain (or anginal equivalent) in a patient without known significant coronary artery disease (CAD) or a history of prior myocardial infarction.
  Interventions: Diagnostic Test: Corus CAD

INTERVENTIONS:
Diagnostic Test: Corus CAD — Age/Sex/Gene Expression Score (ASGES)

SUMMARY:
This is a prospective, multi-center study examining the clinical impact of the Corus CAD (Age/Sex/Gene Expression score - ASGES) assay in approximately 250 evaluable subjects with no history of obstructive coronary artery disease who now present with chest pain or anginal-equivalent symptoms to a primary care physician (PCP) for evaluation.

DETAILED DESCRIPTION:
In symptomatic patients with or without prior cardiac testing, the PCP will initially decide the subject's pretest probability for coronary artery disease (CAD) based on the subject's risk factors and quality of chest pain (typical or atypical), or anginal equivalent (e.g., jaw, arm pain, or unexplained shortness of breath) and consider the results of prior testing, if applicable. The initial questionnaire will capture the PCP's initial clinical impression and decision ('preliminary decision') on how to further evaluate and manage the patient. A Corus CAD (Age/Sex/Gene Expression score - ASGES) assay will be performed at the PCP's office. After the PCP has received the Corus CAD (ASGES) result (approximately 2-3 days later), the PCP will decide on the appropriate evaluation and management of the patient ('final decision') using the Corus CAD (ASGES) result in conjunction with his/her clinical impression and/or other clinical data available. The primary aim of this study is to evaluate whether the Corus CAD (ASGES) test results is associated with a change in the PCPs' diagnostic evaluation and management of patients as compared to their initial testing and treatment decisions.

Since it takes approximately two days for the physician to receive the result of the Corus CAD (ASGES), symptomatic subjects with unstable angina, or suspicion for myocardial infarction will be excluded from the study.

A follow-up phone call and a detailed questionnaire will be performed at 30 + 15 days, from the time of blood draw, to assess the triage decision, such as referral to any subspecialists (cardiologist, gastroenterologist, and pulmonologist), cardiac diagnostic tests performed, cardiac procedures performed, and results of these cardiac tests and procedures.

ELIGIBILITY:
Inclusion Criteria:

1. Stable chest pain, typical or atypical angina or anginal equivalent
2. The patient has signed the appropriate Institutional Review Board approved Informed Consent Form.

Exclusion Criteria:

1. History of myocardial infarction
2. Current Myocardial infarction (MI) or acute coronary syndrome.
3. Current New York Heart Association (NYHA) class III or IV congestive heart failure symptoms.
4. Any previous coronary revascularization.
5. Any individuals with :

   * Diabetes
   * Suspected unstable angina
   * Systemic infections
   * Systemic inflammatory conditions
6. Any individuals currently taking:

   * Steroids
   * Immunosuppressive agents
   * Chemotherapeutic agents
7. Any Major Surgery within 2 months

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a prospective, multi-center study examining the clinical impact of the Corus CAD (Age/Sex/Gene Expression score - ASGES) assay in approximately 250 evaluable subjects with no history of obstructive coronary artery disease who now present with chest pain or anginal-equivalent symptoms to a primary care physician (PCP) for evaluation.
Sampling Method: Probability Sample
Enrollment: 251 (Actual)
Dates: Start 2012-04; Primary Completion 2013-01 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: May Yau, MS, Study Director — CardioDx
Locations (4):
- United States (4):
  - John's Creek Primary Care, Suwanee, Georgia
  - The Lipid Center, Baton Rouge, Louisiana
  - Carolina Family Healthcare, Charlotte, North Carolina
  - Family Care Clinic, Bonham, Texas

REFERENCES:
- [Result] Herman L, Froelich J, Kanelos D, St Amant R, Yau M, Rhees B, Monane M, McPherson J. Utility of a genomic-based, personalized medicine test in patients presenting with symptoms suggesting coronary artery disease. J Am Board Fam Med. 2014 Mar-Apr;27(2):258-67. doi: 10.3122/jabfm.2014.02.130155. PMID 24610188
- [Derived] Ladapo JA, Herman L, Weiner BH, Rhees B, Castle L, Monane M, McPherson JA. Use of a blood test incorporating age, sex, and gene expression influences medical decision-making in the evaluation of women presenting with symptoms suggestive of obstructive coronary artery disease: summary results from two ambulatory care studies in primary care. Menopause. 2015 Nov;22(11):1224-30. doi: 10.1097/GME.0000000000000443. PMID 25828395

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects are enrolled at multiple participating primary care practices from site initiation (Apr-Jun 2012) thru January 2013.
Pre-assignment Details: 327 screened, 275 met inclusion/exclusion. Subjects were excluded from the analysis set if no Corus CAD test could be resulted (7) or if additional information was available and used in making post treatment decisions (3) or did not inclusion/exclusion (discovered after research blood sample draw). Analysis set was 251.
Groups:
- All Subjects With Corus CAD: Subjects are enrolled at multiple participating primary care practices. The main inclusion criterion for enrollment and being tested with Corus CAD is the occurrence of chest pain (or anginal equivalent) in a patient without known significant CAD or a history of prior myocardial infarction.
Period: Overall Study
Arm/Group | All Subjects With Corus CAD
Started | 251
Completed | 249
Not Completed | 2
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Population: Sequentially enrolled subjects meeting the inclusion/exclusion criteria and have a resulted CORUS CAD test.
Groups:
- All Subjects: Subjects are enrolled at multiple participating primary care practices. The main inclusion criterion for enrollment is the occurrence of chest pain (or anginal equivalent) in a patient without known significant CAD or a history of prior myocardial infarction.
Arm/Group | All Subjects
Number analyzed (Participants) | 251
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 182
  >=65 years | 69
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.2 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 140
  Male | 111
Region of Enrollment [Number; unit: participants]
  United States | 251
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 29.7 (6.7)
Age/Sex/Gene Expression Score [Mean (Standard Deviation); unit: unitless] — The ASGES algorithm comprises expression values for 23 genes from peripheral blood cells in 6 terms, patient age, and sex. There are both sex-specific and common algorithm terms with sex-specific weights. The changes in gene expression are quantified using an algorithm that generates a ASGES ranging from 1 to 40. A score less than or equal to 5 indicates a low risk of underlying obstructive coronary disease.The ASGES has been shown to have a negative predictive value of 96% for ASGES less than or equal to 15 in a population referred to MPI.
  unitless | 16 (10)

OUTCOME MEASURES:

1. Primary Outcome: Change in Clinicians' Treatment Decision After Age/Sex/Gene Expression Score
Description: The primary objective was to assess whether the Age/Sex/Gene Expression Score (ASGES) altered clinicians' evaluations, defined by a change in patient management from preliminary to final decision. The change was prospectively defined as a downgrade or upgrade in intensity of the diagnostic plan based on the following hierarchical categories:(1) no further cardiac testing or treatment, (2) lifestyle changes or medical therapy, (3) stress testing (with or without imaging) or computed tomography/coronary angiography, or (4) invasive coronary angiography. The ASGES algorithm comprises expression values for 23 genes from peripheral blood cells in 6 terms, patient age, and sex. The changes in gene expression are quantified using an algorithm that generates a ASGES ranging from 1 to 40. A score <=15 indicates a low risk of underlying obstructive coronary disease. The ASGES has a negative predictive value of 96% for ASGES <=15 in a population referred to myocardial perfusion imaging.
Time Frame: pre- and post- gene expression testing results (on average 2-3 days to receive ASGES)
Population: The study sites included 9 clinicians at 4 community-based primary care practices who assessed all participants with a valid ASGES.
Measure: Number; unit: number of subjects
Groups:
- No Tests/Treatment: Physician decision for no additional tests or cardiac treatment after receiving patients' GES
- Medical Therapy: Physician decision for lifestyle changes or medical therapy after receiving patients' GES
- Stress Test: Physician decision for stress testing (with or without imaging) or computed tomography/coronary angiography after receiving patients' GES
- Invasive Angiography: Physician decision for invasive coronary angiography after receiving patients' GES
Arm/Group | No Tests/Treatment | Medical Therapy | Stress Test | Invasive Angiography
Number analyzed (Participants) | 123 | 22 | 104 | 2
number of subjects
  No Tests/Treatment pre-ASGES, ASGES <=15 (n=40) | 38 | 1 | 1 | 0
  NoTests/Treatment pre-ASGES, ASGES >15 (n=43) | 3 | 1 | 39 | 0
  Medical Therapy pre-ASGES, ASGES ,=15 (n=33) | 25 | 7 | 1 | 0
  Medical Therapy pre-ASGES, ASGES >15 (n=15) | 5 | 2 | 7 | 1
  Stress Tes pre-ASGES, ASGES <=15 (N=53) | 45 | 5 | 3 | 0
  Stress test pre-ASGES, ASGES >15 (n=65) | 5 | 6 | 53 | 1
  Invasive Coronary Angio pre-ASGES, AGES >=15 (n=1) | 1 | 0 | 0 | 0
  Invasive Coronary Angio pre-ASGES, ASGES >15 (n=1) | 1 | 0 | 0 | 0
Statistical Analysis 1: Comparison: No Tests/Treatment; The proportion of patients whose final treatment plan changes from the preliminary will be estimated, and a one-sided binomial test with alpha level of .05 will be used to test whether it is greater than 10%. This is the level at which it is assumed that patient management has been modified by a practically important amount; Test type: Superiority or Other; p < 0.001, one-sided binomial with alpha level of 0

ADVERSE EVENTS:
Arm/Group | All Subjects
Serious Adverse Events (participants affected / at risk) | 0/251
Other Adverse Events (participants affected / at risk) | 0/251

LIMITATIONS AND CAVEATS:
Prospective design may have influenced the diagnostic strategy; but historical controls had a similar diagnostic strategy.

Possible Selection bias; we believe these pts are typical of each practice. Appropriateness of care not evaluated

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
CardioDx will provide a copy of the proposed publication to Collaborator for prior review for a thirty (30)-day period, during which period any Collaborator personnel listed as authors may either (a) elect to opt out from being listed as an author, or (b) suggest modifications to the proposed publication, and if they do not elect either (a) or (b) within that period, they will be deemed to have consented to publication as an author.